CLINICAL TRIAL: NCT07051629
Title: A Phase 1, Double-Blind, Placebo-Controlled, Randomized, Single and Multiple Ascending Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SIF001 in Healthy Subjects and in a Patient Cohort With Epilepsy
Brief Title: Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics And Pharmacodynamics of SIF001 in Healthy Subjects and in Epilepsy Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suninflam Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SIF001-001
Record Dates: First submitted 2025-06-17; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy; Healthy Volunteer
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: The study has two stages. Healthy volunteers in stage 1 of a single ascending dose (SAD) study and in stage 2 of a multiple ascending dose (MAD) study will receive a starting dose of 10mglkg, followed by an ascending dose of 20mg/kg. A cohort of epilepsy patients will be added to stage 2.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SIF001 10-20mg/kg IV (Experimental): SIF001 infused intravenously over one hour
  Interventions: Biological: SIF001
- Placebo (Placebo Comparator): Placebo infused intravenously over one hour
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: SIF001 — SIF001 intravenous infusion every two weeks
  Arms: SIF001 10-20mg/kg IV
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a dose escalation study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of SIF001, a monoclonal antibody with the potential to treat epilespy

DETAILED DESCRIPTION:
Nonclinical studies including disease animal model studies and toxicological studies indicate that SIF001 has the potential to be a therapeutical agent for epilepsy treatment through addressing the underlying pathology. This a phase 1 dose escalation study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of SIF001 in healthy subjects and in a patient cohort with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

-

Healthy Volunteers Only (Stage I and II (Phase 1a and 1b)):

1. Male or female 18 to 55 years of age at the time of signing the informed consent.
2. In good health as determined by the Investigator, based on medical history and screening evaluations.
3. Body weight of ≥ 50 kg and BMI within the range 18-30 kg/m2 (inclusive)

   Patients with Epilepsy Only (Stage II (Phase 1b)):
4. Male or female 18 to 70 years of age at the time of signing the informed consent.
5. A clinical diagnosis of focal or generalized epilepsy. Subjects must have motor seizures, with or without impaired awareness.
6. Has a minimum of 4 seizures per 4-week period while taking 1 to 3 anti-seizure medications
7. All medications and epilepsy interventions must be stable for 8 weeks before screening and are expected to remain stable during the study

   All Subjects:
8. Negative serum pregnancy test at screening and urine pregnancy test on Day -1 before starting study treatment in all pre-menopausal women and women < 12 months after the onset of menopause.
9. Female participants of child-bearing potential and male participants must agree to use adequate contraception for the duration of the protocol.
10. Able to sign informed consent and comply with the protocol.

Exclusion Criteria:

* Healthy Volunteers (Stage I and II (Phase 1a and 1b)):

  1. Subjects with any unresolved history of clinically significant disease, in the opinion of the investigator.
  2. Past or intended use of over-the-counter (OTC) or prescription medication (other than ≤ 2 g/day paracetamol [acetaminophen] or ≤ 800-mg/day ibuprofen), vitamins, and dietary or herbal supplements within 7 days or 5 half-lives of the respective drug, if known (whichever is longer), prior to dosing.

     Patients with Epilepsy (Stage II (Phase 1b)):
  3. Acute precipitant of seizure within the past 3 months prior to screening such as major trauma, hypoglycemia, hyperglycemia, cardiac arrest, or post-anoxia

     All Subjects:
  4. Any uncontrolled medical or psychiatric condition (e.g., hypertension, diabetes, chronic obstructive pulmonary disorder, asthma, depression) as judged by the investigator.
  5. Any clinically significant findings in medical examination, including physical examination, 12-lead ECG, vital signs, clinical laboratory tests. Specifically:

     1. alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 × upper limit of normal (ULN), Total bilirubin ≥ 2 × ULN
     2. QT interval corrected by Fridericia's formula (QTcF) > 450 msec (male) or > 470 msec (female)
  6. Undergone major surgery ≤ 2 months prior to Day -1.
  7. Received any investigational drug within 30 days or 5 half-lives (whichever is longer, if known) before screening.
  8. Received any vaccine within 6 weeks before planned SIF001 administration.
  9. Loss of more than 100 mL blood (e.g., a blood donation) within 2 months before Day -1, or has received any blood, plasma, or platelet transfusions within 3 months before admission.
  10. Active liver disease or severe renal impairment, including serum creatinine ≥ 1.5 × ULN or estimated glomerular filtration rate of < 60 mL/min/1.73m2.
  11. Known history of substance use disorder.
  12. History of active human immunodeficiency virus (HIV), active hepatitis C virus (HCV), or active hepatitis B virus (HBV)
  13. Recent (2 weeks) history of a positive COVID-19 test result or disease symptoms of COVID-19 disease such as shortness of breath, cough, rhinorrhea, sore throat etc.
  14. Known history of hypersensitivity or anaphylactic reaction to intravenous medications, biologicals, or fluids.
  15. History of any clinically significant disease or disorder which, in the opinion of the investigators, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
  16. History of status epilepticus within 2 years of screening
  17. Known history of suicidality within 2 years of screening, or answering "yes" to questions 4 and 5 of the Columbia Suicide Severity Rating Scale (C-SSRS)
  18. Unable to complete this study for other reasons or the investigator believes that the subject should be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants and rate of treatment-related adverse events assessed by dose group and by active treatment vs placebo | Day 1 to Day 15 for SAD, and Day 1 to Day 43 for MAD
  To measure the incidence and severity of adverse events (AEs) and severe adverse events (SAEs), clinical laboratory parameters, vital signs, and physical examinations,

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters/ profiles:Area under the plasma concentration versus time curve (AUC) | Through Day 75
  PK: AUC D0-∞
Pharmacokinetic (PK) profile/parameters: Maximum observed plasma concentration | Through Day 75
  PK: Cmax
Pharmacokinetic (PK) profile/parameters: Time at which maximum plasma concentration occurs | Through Day 75
  PK: tmax
Pharmacokinetic (PK) profile/parameters: terminal elimination phase half life | Through Day 75
  PK: t(1/2)
Pharmacokinetic (PK) profile/parameters: total clearance | Through Day 75
  PK: CL
Pharmacokinetic (PK) profile/parameters: volume of distribution | Through Day 75
  PK: Vd
Incidence of immunogenicity of SIF001 (production of anti-SIF001 antibodies) | Through Day 75
  Detection of anti-SIF001 antibodies
To evaluate the change from baseline in seizure frequency (patient cohort only) | from Day 1 to 29 (4 weeks), from Day 29 to 57 (4 weeks), and up to Day 57 in patients with epilepsy
  Frequency of observed countable seizures with motor manifestations, with or without impaired awareness

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Accel Research sites network, DeLand, Florida
  - Quest Research Institute, Farmington Hills, Michigan

IPD SHARING:
Plan to Share IPD: No